CLINICAL TRIAL: NCT00039442
Title: A Phase II Evaluation Of Capecitabine (NSC #712807) In The Treatment Of Persistent Or Recurrent Non-Squamous Cell Carcinoma Of The Cervix
Brief Title: Capecitabine in Treating Patients With Persistent or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0128G; NCI-2012-02469 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000069384; GOG-0128G (Other: Gynecologic Oncology Group); GOG-0128G (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Recurrent Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Capecitabine

ARMS (1):
- Treatment (Experimental): Patients receive oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Capecitabine — Given orally
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of capecitabine in treating patients who have persistent or recurrent cervical cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor activity of capecitabine in patients with persistent or recurrent non-squamous cell carcinoma of the cervix who have failed higher priority treatment protocols.

II. Determine the nature and degree of toxicity of this drug in these patients. III. Determine whether the mRNA tumor expression levels of thymidylate synthase (TS), dihydropyrimidine dehydrogenase (DPD), and thymidine phosphorylase (TP) at baseline are potential predictors of clinical outcomes (response and survival) in patients treated with this drug.

IV. Determine whether the serum level of TP is a potential prognostic indicator of clinical outcomes (response and survival) in patients treated with this drug.

V. Determine whether the TS promoter polymorphism in peripheral blood is a potential prognostic indicator of clinical outcomes (response and survival) in patients treated with this drug.

VI. Determine the associations among the various measures of TS, DPD, and TP and clinical outcomes (response and survival) in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary non-squamous cell carcinoma (non-SCC) of the cervix

  * Persistent or recurrent disease
  * Eligible subtypes include:

    * Adenocarcinoma
    * Adenosquamous cell carcinoma
    * Undifferentiated carcinoma
* Documented disease progression
* At least 1 unidimensionally measurable target lesion outside prior irradiation field

  * At least 20 mm by conventional techniques (e.g., palpation, plain x-ray, CT scan, and MRI)
  * At least 10 mm by spiral CT scan
* Received 1 prior systemic chemotherapy regimen for advanced, metastatic, or recurrent non-SCC of the cervix

  * Radiosensitizing chemotherapy administered in combination with primary radiotherapy is not counted as a systemic chemotherapy regimen
* Tissue blocks from initial diagnosis, metastasis, or recurrence available for submission to the GOG tissue bank
* Ineligible for higher priority Gynecologic Oncology Group (GOG) protocol (if one exists), defined as any Temporarily closed GOG phase III protocol for the same patient population
* Performance status - GOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine clearance at least 50 mL/min
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No Temporarily closed infection requiring antibiotics
* No grade 2 or greater sensory or motor neuropathy
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* At least 3 weeks since prior biological or immunological anticancer agents
* No more than 1 prior non-cytotoxic biologic therapy or cytostatic regimen (e.g., monoclonal antibodies, cytokines, or small-molecule inhibitors of signal transduction) for recurrent or persistent non-SCC of the cervix
* See Disease Characteristics
* See Biologic therapy
* At least 3 weeks since prior chemotherapy and recovered
* No prior capecitabine
* No more than 1 prior cytotoxic chemotherapy regimen (either with single or combination cytotoxic drug therapy)
* At least 1 week since prior hormonal anticancer therapy
* Concurrent hormone replacement therapy allowed
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* Recovered from prior recent surgery
* At least 3 weeks since other prior anticancer therapy
* No prior cancer treatment that would preclude this study therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2002-04-29 (Actual); Primary Completion 2005-12-07 (Actual)

PRIMARY OUTCOMES:
Duration of objective response | Up to 7 years
Frequency of adverse events, graded according to CTC version 2.0 | Up to 7 years
Frequency of objective response | Up to 7 years
Severity of observed adverse events, graded according CTC version 2.0 | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Look, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group of Arizona, Phoenix, Arizona, United States